CLINICAL TRIAL: NCT04490018
Title: Immunogenicity and Safety Study of a Quadrivalent Meningococcal Conjugate Vaccine Versus Nimenrix®, and When Administered Alone or Concomitantly With 9vHPV and Tdap-IPV Vaccines in Healthy Adolescents
Brief Title: Study on a Quadrivalent Meningococcal Conjugate Vaccine (MenACYW Conjugate Vaccine) Compared to a Meningococcal Reference Vaccine, and When Given Alone or With Two Other Vaccines in Healthy Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEQ00071; 2020-001665-37 (EudraCT Number); U1111-1249-2973 (Registry Identifier: ICTRP)
Record Dates: First submitted 2020-07-27; First posted 2020-07-28 (Actual); Results first posted 2023-06-06 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Meningococcal Immunisation; Healthy Volunteers
MeSH Terms: interventions — Tetanus Toxoid; Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Intervention Model Description: This was a parallel group prevention study with 2 groups that were observer blind (only the person administering the vaccine was unblinded), and 1 group that was open-label.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study was performed in a partially observer-blind fashion:
  In Groups 1 and 2
  * Investigators and study staff who conducted the safety assessment, participants, parents/legally acceptable representatives, the Sponsor, and laboratory personnel performing the serology testing were kept blinded to the vaccine received.
  * Only the study staff who prepared and administered the vaccine and were not involved with the safety evaluation know which vaccine was administered.
  In Group 3
  - Everyone involved in the study (i.e., Investigator, study staff, the Sponsor, participants, parents/legally acceptable representatives) know which vaccine was administered. This open-label design for Group 3 was due to the different vaccination schedule for this group than for Groups 1 and 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) (Experimental): Participants received 0.5-milliliter (mL) intramuscular injection of MenACYW Conjugate vaccine on Day 01 and 0.5-mL intramuscular injection of 9vHPV + Tdap-IPV vaccines (sequentially after MenACYW vaccine) at Day 31.
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine (MenACYW Conjugate vaccine); Biological: Human Papillomavirus 9-valent Vaccine (9vHPV); Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed Combined with Inactivated Poliomyelitis Vaccine (Tdap-IPV)
- Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) (Active Comparator): Participants received 0.5-mL intramuscular injection of Nimenrix® vaccine on Day 01 and 0.5-mL intramuscular injection of 9vHPV + Tdap-IPV vaccines (sequentially after Nimenrix® vaccine) at Day 31.
  Interventions: Biological: Meningococcal group A, C, W-135, and Y conjugate vaccine; Biological: Human Papillomavirus 9-valent Vaccine (9vHPV); Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed Combined with Inactivated Poliomyelitis Vaccine (Tdap-IPV)
- Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration) (Experimental): Participants received 0.5-mL intramuscular injection of MenACYW Conjugate vaccine concomitantly with 9vHPV + Tdap-IPV vaccines on Day 01.
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine (MenACYW Conjugate vaccine); Biological: Human Papillomavirus 9-valent Vaccine (9vHPV); Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed Combined with Inactivated Poliomyelitis Vaccine (Tdap-IPV)

INTERVENTIONS:
Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine (MenACYW Conjugate vaccine) — Pharmaceutical form: Liquid solution for injection Route of administration: Intramuscular
  Other Names: MenQuadfi®
  Arms: Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration); Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration)
Biological: Meningococcal group A, C, W-135, and Y conjugate vaccine — Pharmaceutical form: Powder and solvent for solution for injection Route of administration: Intramuscular
  Other Names: Nimenrix®
  Arms: Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration)
Biological: Human Papillomavirus 9-valent Vaccine (9vHPV) — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
  Other Names: Gardasil® 9
Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed Combined with Inactivated Poliomyelitis Vaccine (Tdap-IPV) — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
  Other Names: Repevax®/Triaxis®/Adacel®Polio

SUMMARY:
Primary Objective:

To demonstrate the non-inferiority of the seroprotection rate (serum bactericidal assay using human complement [hSBA] titer greater than or equal to [>=] 1:8) to meningococcal serogroups A, C, W, and Y following the administration of a single dose of Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate vaccine (MenACYW Conjugate vaccine) (Group 1) compared to a single dose of Nimenrix® (Group 2).

Secondary Objective:

To describe:

* the antibody response of meningococcal serogroups A, C, W, and Y measured by hSBA, before and 1 month following meningococcal vaccination administered alone (Groups 1 and 2) or concomitantly with 9-valent human papilloma virus (9vHPV) and tetanus, diphtheria, and acellular pertussis - inactivated polio vaccine [adsorbed, reduced antigen(s) content] (Tdap-IPV) vaccines (Group 3).
* the antibody response of meningococcal serogroup C measured by hSBA and serum bactericidal assay using baby rabbit complement (rSBA), before vaccination and at Day 31 after vaccination with MenACYW Conjugate vaccine or Nimenrix® (Groups 1 and 2) according to MenC primed status.
* the antibody response against antigens of 9vHPV and Tdap-IPV vaccines, before and 1 month following vaccination.
* the safety profile in each group after each and any vaccination.

DETAILED DESCRIPTION:
The duration of study participation for each participant was approximately 30 to 60 days, including 2 or 3 visits (1 or 2 vaccination visit) and 1 or 2 telephone calls, depending on study Group.

* This was the first dose of 9vHPV, of the 2-dose or 3-dose series according to the local recommendations and age of the participant. These additional vaccinations for the completion of 9vHPV schedule took place outside of the objectives and scope of this study and thus were not described in this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Aged 10 to 17 years on the day of inclusion ('10 to 17 years' means from the day of the 10th birthday to the day before the 18th birthday).
* Meningococcal serogroup C Conjugate vaccine (MenC) naïve participants or participants having received monovalent MenC priming in infancy (less than [<] 2 years of age).
* Assent form had been signed and dated by the participant as per local regulation, and Informed Consent Form had been signed and dated by the parent/legally acceptable representative and by the participant if she/he turns 18 years old during the study.
* Participants and parent/legally acceptable representative were able to attend all scheduled visits and compiled with all study procedures.
* Covered by health insurance, if required by local regulations.

Exclusion Criteria:

* Participant was pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after last vaccination. To be considered of non-childbearing potential, a female must be pre-menarche.
* Previous vaccination against meningococcal disease with either the study vaccine or another vaccine (i.e., polysaccharide, or conjugate meningococcal vaccine containing serogroups A, C, W, or Y; or meningococcal B serogroup-containing vaccine), except licensed monovalent MenC vaccination received before 2 years of age.
* Participation at the time of study enrollment (or in the 4 weeks preceding the first study vaccination) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks preceding any study vaccination or planned receipt of any vaccine in the 4 weeks following any study vaccination except for influenza vaccination, which might receive at least 2 weeks before study vaccines. This exception included monovalent pandemic influenza vaccines and multivalent influenza vaccines.
* History of vaccination with any tetanus, diphtheria, pertussis, or inactivated polio virus vaccine within the previous 3 years.
* Previous human papilloma virus (HPV) vaccination.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* History of meningococcal infection, confirmed either clinically, serologically, or microbiologically.
* Known history of diphtheria, tetanus, pertussis, poliomyelitis, and/or HPV infection or disease.
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the study or to a vaccine containing any of the same substances.
* Personal history of Guillain-Barré syndrome.
* Personal history of an Arthus-like reaction after vaccination with a tetanus toxoid-containing vaccine within at least 10 years of the proposed study vaccination.
* Personal history of new or past encephalopathy, progressive or unstable neurological disorder, or unstable epilepsy.
* Verbal report of thrombocytopenia, contraindicating intramuscular vaccination.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction.
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with study conduct or completion.
* Moderate or severe acute illness/infection (according to Investigator's judgment) on the day of vaccination or febrile illness (temperature >= 38.0 degree Celsius [>= 100.4 degree Fahrenheit]). A prospective participant should not be included in the study until the condition had resolved or the febrile event has subsided.
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.
* Participant at high risk for meningococcal infection during the study (specifically but not limited to participants with persistent complement deficiency, with anatomic or functional asplenia, or participants traveling to countries with high endemic or epidemic disease.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 463 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (23):
- Hungary (5):
  - Investigational Site Number :3480003, Budapest
  - Investigational Site Number :3480001, Győr
  - Investigational Site Number :3480002, Miskolc
  - Investigational Site Number :3480004, Szigetvár
  - Investigational Site Number :3480006, Szombathely
- Italy (5):
  - Investigational Site Number :3800005, Foggia, Apulia
  - Investigational Site Number :3800006, Catanzaro, Calabria
  - Investigational Site Number :3800002, Milan, Lombardy
  - Investigational Site Number :3800004, Palermo, Sicily
  - Investigational Site Number :3800001, Genova
- Investigational Site Number :7020002, Singapore, Singapore
- Spain (12):
  - Investigational Site Number :7240001, Seville, Andalusia
  - Investigational Site Number :7240002, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number :7240005, Esplugues de Llobregat, Castille and León
  - Investigational Site Number :7240006, Santiago de Compostela, Galicia [Galicia]
  - Investigational Site Number :7240003, Madrid, Madrid, Comunidad de
  - Investigational Site Number :7240011, Burriana, Valenciana, Comunidad
  - Investigational Site Number :7240007, Puçol, Valenciana, Comunidad
  - Investigational Site Number :7240008, Valencia, Valenciana, Comunidad
  - Investigational Site Number :7240004, Valencia, Valenciana, Comunidad
  - Investigational Site Number :7240009, Valencia, Valenciana, Comunidad
  - Investigational Site Number :7240010, Valencia, Valenciana, Comunidad
  - Investigational Site Number :7240012, Valencia, Valenciana, Comunidad

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Diez-Domingo J, Simko R, Icardi G, Chong CP, Zocchetti C, Syrkina O, Bchir S, Bertrand-Gerentes I. Immunogenicity and Safety of a Quadrivalent Meningococcal Conjugate Vaccine Versus Nimenrix in Healthy Adolescents: A Randomized Phase IIIb Multicenter Study. Infect Dis Ther. 2024 Aug;13(8):1835-1859. doi: 10.1007/s40121-024-01009-x. Epub 2024 Jul 2. PMID 38955966
- See also: MEQ00071 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25311&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 21 active centers in Hungary, Italy, Spain and Singapore between 16 March 2021 to 11 May 2022.
Pre-assignment Details: A total of 463 participants were enrolled and randomized in this study.
Groups:
- Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration): Participants received 0.5 milliliters (mL) intramuscular injection of Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate vaccine (MenACYW Conjugate vaccine) on Day 01 and 0.5-mL intramuscular injection of 9-valent human papilloma virus (9vHPV) + tetanus, diphtheria, and acellular pertussis - inactivated polio vaccines (Tdap-IPV) (sequentially after MenACYW vaccine) at Day 31.
- Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration): Participants received 0.5 mL intramuscular injection of Nimenrix® vaccine on Day 01 and 0.5-mL intramuscular injection of 9vHPV + Tdap-IPV vaccines (sequentially after Nimenrix® vaccine) at Day 31.
- Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration): Participants received 0.5 mL intramuscular injection of MenACYW Conjugate vaccine concomitantly with 9vHPV + Tdap-IPV vaccines on Day 01.
Period: Overall Study
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration)
Started | 173 | 173 | 117
Safety Analysis Set (Participants who had received at least one dose of the study vaccines (all groups) and had any safety data available.) | 171 | 171 | 116
Vaccinated at Day 01 | 170 | 172 | 116
Vaccinated at Day 31 | 168 | 169 | 0 (Group 3 participants did not receive any vaccination at Day 31.)
Completed | 167 | 165 | 116
Not Completed | 6 | 8 | 1
Not completed — Protocol Violation | 0 | 2 | 1
Not completed — Lost to Follow-up | 2 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — Withdrawal by parent/guardian | 2 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration): Participants received 0.5 mL intramuscular injection of MenACYW Conjugate vaccine on Day 01 and 0.5-mL intramuscular injection of 9vHPV + Tdap-IPV vaccines (sequentially after MenACYW vaccine) at Day 31.
- Total: Total of all reporting groups
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration) | Total
Number analyzed (Participants) | 173 | 173 | 117 | 463
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.4 (2.32) | 12.8 (2.38) | 12.5 (2.47) | 12.6 (2.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 57 | 45 | 151
  Male | 124 | 116 | 72 | 312
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 3
  Asian | 2 | 2 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 5
  White | 165 | 169 | 115 | 449
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Antibody Titers >=1:8 Against Meningococcal Serogroups A, C, W, and Y Measured by hSBA Following Vaccination With MenACYW Conjugate Vaccine or Nimenrix® Vaccine (Non-inferiority Analysis): Groups 1 and 2
Description: Antibody titers against meningococcal serogroups A, C, W, and Y were measured by serum bactericidal assay using human complement (hSBA). Non-inferiority data analysis for this outcome measure was planned to be conducted only for Groups 1 and 2, not for Group 3. Group 3 data is reported separately.
Time Frame: Day 31 (post-vaccination)
Population: Analysis was performed on hSBA Per-Protocol Analysis Set for meningococcal vaccines (PPASM) which was a subset that included all participants who received a dose of the study vaccine and had a valid post-vaccination serology result. The participants who presented protocol deviations were excluded from PPASM. Here, 'number analyzed'=participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration)
Number analyzed (Participants) | 159 | 161
percentage of participants
  Serogroup A: number analyzed (Participants) | 159 | 160
  Serogroup A | 97.5 [93.7 to 99.3] | 92.5 [87.3 to 96.1]
  Serogroup C | 100 [97.7 to 100] | 95.0 [90.4 to 97.8]
  Serogroup W | 100 [97.7 to 100] | 98.8 [95.6 to 99.8]
  Serogroup Y: number analyzed (Participants) | 158 | 160
  Serogroup Y | 99.4 [96.5 to 100] | 98.1 [94.6 to 99.6]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) vs Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration); Serogroup A; Test type: Non-Inferiority — The two-sided 95 percent (%) confidence interval (CI) was calculated based on the Wilson score method without continuity correction. The non-inferiority was demonstrated if the lower limit of the 95% CI of the percentage difference between compared groups was greater than (>) -10%; Difference in Percentage = 4.98, 95% CI 2-sided [0.06 to 10.36]
Statistical Analysis 2: Comparison: Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) vs Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration); Serogroup C; Test type: Non-Inferiority — The two-sided 95% CI was calculated based on the Wilson score method without continuity correction. The non-inferiority was demonstrated if the lower limit of the 95% CI of the percentage difference between compared groups was greater > -10%; Difference in Percentage = 4.97, 95% CI 2-sided [1.58 to 9.50]
Statistical Analysis 3: Comparison: Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) vs Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration); Serogroup W; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in Percentage = 1.24, 95% CI 2-sided [-1.28 to 4.42]
Statistical Analysis 4: Comparison: Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) vs Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration); Serogroup Y; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in Percentage = 1.24, 95% CI 2-sided [-1.88 to 4.77]

2. Secondary Outcome: Geometric Mean Titers (GMTs) of Antibodies Measured by hSBA Against Meningococcal Serogroups A, C, Y, and W
Description: GMTs against Meningococcal Serogroups A, C, Y, and W were measured by hSBA. Titers were expressed in terms of 1/dilution.
Time Frame: Day 01 (pre-vaccination) and Day 31 (post-vaccination)
Population: Analysis was performed on hSBA PPASM. Here, 'number analyzed'=participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration)
Number analyzed (Participants) | 159 | 161 | 113
titers
  Serogroup A: Day 01: number analyzed (Participants) | 158 | 160 | 112
  Serogroup A: Day 01 | 6.95 [6.18 to 7.83] | 6.41 [5.67 to 7.26] | 7.38 [6.23 to 8.75]
  Serogroup A: Day 31: number analyzed (Participants) | 159 | 160 | 113
  Serogroup A: Day 31 | 78.2 [64.6 to 94.7] | 56.0 [44.0 to 71.2] | 42.2 [32.5 to 54.7]
  Serogroup C: Day 01: number analyzed (Participants) | 158 | 160 | 113
  Serogroup C: Day 01 | 6.40 [5.17 to 7.92] | 5.51 [4.59 to 6.62] | 5.67 [4.51 to 7.14]
  Serogroup C: Day 31 | 2294 [1675 to 3142] | 619 [411 to 931] | 1938 [1365 to 2752]
  Serogroup Y: Day 01 | 2.56 [2.27 to 2.89] | 3.14 [2.63 to 3.75] | 2.43 [2.09 to 2.84]
  Serogroup Y: Day 31: number analyzed (Participants) | 158 | 160 | 113
  Serogroup Y: Day 31 | 169 [141 to 202] | 84.8 [68.3 to 105] | 171 [138 to 211]
  Serogroup W: Day 01: number analyzed (Participants) | 159 | 161 | 112
  Serogroup W: Day 01 | 3.76 [3.22 to 4.40] | 4.36 [3.68 to 5.17] | 3.98 [3.18 to 4.96]
  Serogroup W: Day 31 | 134 [109 to 164] | 64.6 [52.5 to 79.4] | 74.6 [61.8 to 90.1]

3. Secondary Outcome: Percentage of Participants With hSBA Antibody Titers >=1:4 and >=1:8 Against Meningococcal Serogroups A, C, Y, and W
Description: Antibody titers against Meningococcal Serogroups A, C, Y and W were measured by hSBA. Percentage of participants With hSBA antibody titers >=1:4 and >=1:8 for serogroups A, C, Y, and W were reported in the outcome measure.
Time Frame: Day 01 (pre-vaccination) and Day 31 (post-vaccination)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration)
Number analyzed (Participants) | 159 | 161 | 113
percentage of participants
  Serogroup A: >= 1:4: Day 01: number analyzed (Participants) | 158 | 160 | 112
  Serogroup A: >= 1:4: Day 01 | 94.3 [89.5 to 97.4] | 88.1 [82.1 to 92.7] | 83.9 [75.8 to 90.2]
  Serogroup A: >= 1:8: Day 01: number analyzed (Participants) | 158 | 160 | 112
  Serogroup A: >= 1:8: Day 01 | 56.3 [48.2 to 64.2] | 50.6 [42.6 to 58.6] | 58.9 [49.2 to 68.1]
  Serogroup A: >= 1:4: Day 31: number analyzed (Participants) | 159 | 160 | 113
  Serogroup A: >= 1:4: Day 31 | 98.7 [95.5 to 99.8] | 95.0 [90.4 to 97.8] | 96.5 [91.2 to 99.0]
  Serogroup A: >= 1:8: Day 31: number analyzed (Participants) | 159 | 160 | 113
  Serogroup A: >= 1:8: Day 31 | 97.5 [93.7 to 99.3] | 92.5 [87.3 to 96.1] | 91.2 [84.3 to 95.7]
  Serogroup C: >= 1:4: Day 01: number analyzed (Participants) | 158 | 160 | 113
  Serogroup C: >= 1:4: Day 01 | 61.4 [53.3 to 69.0] | 61.3 [53.2 to 68.8] | 57.5 [47.9 to 66.8]
  Serogroup C: >= 1:8: Day 01: number analyzed (Participants) | 158 | 160 | 113
  Serogroup C: >= 1:8: Day 01 | 41.1 [33.4 to 49.2] | 35.6 [28.2 to 43.6] | 41.6 [32.4 to 51.2]
  Serogroup C: >= 1:4: Day 31 | 100 [97.7 to 100] | 96.3 [92.1 to 98.6] | 99.1 [95.2 to 100]
  Serogroup C: >= 1:8: Day 31 | 100 [97.7 to 100] | 95.0 [90.4 to 97.8] | 99.1 [95.2 to 100]
  Serogroup Y: >= 1:4: Day 01 | 14.5 [9.4 to 20.9] | 17.4 [11.9 to 24.1] | 8.8 [4.3 to 15.7]
  Serogroup Y: >= 1:8: Day 01 | 9.4 [5.4 to 15.1] | 15.5 [10.3 to 22.1] | 6.2 [2.5 to 12.3]
  Serogroup Y: >= 1:4: Day 31: number analyzed (Participants) | 158 | 160 | 113
  Serogroup Y: >= 1:4: Day 31 | 99.4 [96.5 to 100] | 98.8 [95.6 to 99.8] | 100 [96.8 to 100]
  Serogroup Y: >= 1:8: Day 31: number analyzed (Participants) | 158 | 160 | 113
  Serogroup Y: >= 1:8: Day 31 | 99.4 [96.5 to 100] | 98.1 [94.6 to 99.6] | 100 [96.8 to 100]
  Serogroup W: >= 1:4: Day 01: number analyzed (Participants) | 159 | 161 | 112
  Serogroup W: >= 1:4: Day 01 | 39.6 [32.0 to 47.7] | 46.6 [38.7 to 54.6] | 30.4 [22.0 to 39.8]
  Serogroup W: >= 1:8: Day 01: number analyzed (Participants) | 159 | 161 | 112
  Serogroup W: >= 1:8: Day 01 | 22.6 [16.4 to 29.9] | 28.6 [21.7 to 36.2] | 26.8 [18.9 to 36.0]
  Serogroup W: >= 1:4: Day 31 | 100 [97.7 to 100] | 98.8 [95.6 to 99.8] | 100 [96.8 to 100]
  Serogroup W: >= 1:8: Day 31 | 100 [97.7 to 100] | 98.8 [95.6 to 99.8] | 99.1 [95.2 to 100]

4. Secondary Outcome: Percentage of Participants With >= 4-Fold Rise In hSBA Antibody Titers Against Meningococcal Serogroups A, C, Y, and W
Description: Antibody titers against Meningococcal Serogroups A, C, Y and W were measured by hSBA. Fold-rise was calculated as ratio of post-dose titer on Day 31 to pre-dose titer on Day 01.
Time Frame: From Baseline (Day 01) to Day 31 (post-vaccination)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration)
Number analyzed (Participants) | 159 | 161 | 113
percentage of participants
  Serogroup A: number analyzed (Participants) | 158 | 159 | 112
  Serogroup A | 88.0 [81.9 to 92.6] | 76.1 [68.7 to 82.5] | 65.2 [55.6 to 73.9]
  Serogroup C: number analyzed (Participants) | 158 | 160 | 113
  Serogroup C | 99.4 [96.5 to 100] | 91.9 [86.5 to 95.6] | 97.3 [92.4 to 99.4]
  Serogroup Y: number analyzed (Participants) | 158 | 160 | 113
  Serogroup Y | 98.7 [95.5 to 99.8] | 92.5 [87.3 to 96.1] | 99.1 [95.2 to 100]
  Serogroup W: number analyzed (Participants) | 159 | 161 | 112
  Serogroup W | 94.3 [89.5 to 97.4] | 88.2 [82.2 to 92.7] | 86.6 [78.9 to 92.3]

5. Secondary Outcome: Percentage of Participants With Vaccine Seroresponse Against Meningococcal Serogroups A, C, Y, and W
Description: Antibody titers against meningococcal serogroups A, C, Y, and W were measured by hSBA. The vaccine seroresponse was defined as a post-vaccination hSBA titer greater than or equal to (>=) 1:16 for participants with pre-vaccination hSBA titer less than (<) 1:8, or a >= 4-fold increase in hSBA titer from pre-vaccination to post-vaccination for participants with pre-vaccination hSBA titer >= 1:8.
Time Frame: Day 31 (post-vaccination)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration)
Number analyzed (Participants) | 159 | 161 | 113
percentage of participants
  Serogroup A: number analyzed (Participants) | 158 | 159 | 112
  Serogroup A | 88.0 [81.9 to 92.6] | 75.5 [68.0 to 81.9] | 63.4 [53.8 to 72.3]
  Serogroup C: number analyzed (Participants) | 158 | 160 | 113
  Serogroup C | 99.4 [96.5 to 100] | 88.8 [82.8 to 93.2] | 97.3 [92.4 to 99.4]
  Serogroup Y: number analyzed (Participants) | 158 | 160 | 113
  Serogroup Y | 98.7 [95.5 to 99.8] | 88.1 [82.1 to 92.7] | 99.1 [95.2 to 100]
  Serogroup W: number analyzed (Participants) | 159 | 161 | 112
  Serogroup W | 93.1 [88.0 to 96.5] | 81.4 [74.5 to 87.1] | 85.7 [77.8 to 91.6]

6. Secondary Outcome: Geometric Mean Titers (GMTs) of Antibodies Measured by hSBA Against Meningococcal Serogroup C: Meningococcal Serogroup C Conjugate Vaccine (MenC) Primed Participants in Groups 1 and 2
Description: GMTs against meningococcal Serogroup C in MenC primed participants (participants who received monovalent MenC priming in infancy < 2 years of age) were measured by hSBA. Titers were expressed in terms of 1/dilution.
Time Frame: Day 01 (pre-vaccination) and Day 31 (post-vaccination)
Population: Analysis was performed on participants who were MenC primed, received a dose of the study vaccine and had a valid post-vaccination serology result. The participants who presented protocol deviations were excluded. Here, 'number analyzed' = participants with available data for specified category. Data for this outcome measure was not planned to be collected and analyzed for Group 3.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration)
Number analyzed (Participants) | 114 | 112
titers
  Day 01: number analyzed (Participants) | 113 | 111
  Day 01 | 7.30 [5.64 to 9.45] | 7.06 [5.57 to 8.95]
  Day 31 | 4222 [3166 to 5632] | 2361 [1740 to 3204]

7. Secondary Outcome: Geometric Mean Titers (GMTs) of Antibodies Measured by Serum Bactericidal Assay Using Baby Rabbit Complement (rSBA) Against Meningococcal Serogroups C: Meningococcal Serogroup C Conjugate Vaccine (MenC) Primed Participants in Groups 1 and 2
Description: GMTs against Serogroup C in MenC primed participants (participants who received monovalent MenC priming in infancy < 2 years of age) were measured by rSBA. Titers were expressed in terms of 1/dilution.
Time Frame: Day 01 (pre-vaccination) and Day 31 (post-vaccination)
Population: Analysis was performed on participants who were MenC primed. Here, "overall number of participants analyzed" signifies participants with available data for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for Group 3.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration)
Number analyzed (Participants) | 37 | 37
titers
  Day 01 | 6.51 [3.56 to 11.9] | 3.32 [2.24 to 4.91]
  Day 31 | 19760 [13308 to 29338] | 7052 [4706 to 10567]

8. Secondary Outcome: Geometric Mean Concentrations (GMCs) of Anti-Diphtheria, Tetanus Antibodies Contained in Tetanus, Diphtheria, and Acellular Pertussis - Inactivated Polio Vaccine (Tdap-IPV) Vaccine in Groups 1 and 2
Description: Geometric mean concentrations of anti-Diphtheria, and tetanus antibodies were measured by electro chemiluminescent method. Blood samples were assessed for participants at Day 31 and at Day 61, respectively.
Time Frame: Day 31 (post-vaccination) and Day 61 (post-vaccination)
Population: Analysis performed on Per-Protocol Analysis Set for concomitant vaccines (PPASC) which was a subset that included all participants who received a dose of study vaccine and had a valid post-vaccination serology result. Participants who presented protocol deviations and who did not produce a valid test result were excluded from PPASC. Here, 'number analyzed'=participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: International units/milliliter (IU/mL)
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration)
Number analyzed (Participants) | 149 | 147
International units/milliliter (IU/mL)
  Anti-Tetanus: Day 31: number analyzed (Participants) | 147 | 147
  Anti-Tetanus: Day 31 | 25.5 [22.0 to 29.5] | 18.4 [15.8 to 21.5]
  Anti-Tetanus: Day 61 | 17.3 [14.9 to 20.1] | 16.1 [14.1 to 18.5]
  Anti-Diphteria: Day 31: number analyzed (Participants) | 147 | 147
  Anti-Diphteria: Day 31 | 0.200 [0.169 to 0.238] | 0.215 [0.181 to 0.254]
  Anti-Diphteria: Day 61 | 3.75 [3.24 to 4.35] | 3.88 [3.37 to 4.47]

9. Secondary Outcome: Geometric Mean Concentrations (GMCs) of Anti-Polio Antibodies Contained in Tetanus, Diphtheria, and Acellular Pertussis - Inactivated Polio Vaccine (Tdap-IPV) Vaccine in Groups 1 and 2
Description: GMCs of anti-poliovirus types 1, 2, and 3 were measured by neutralization assay. Concentrations were expressed in terms of titers (1/dilution). Blood samples were assessed for participants at Day 31 and at Day 61, respectively.
Time Frame: Day 31 (post-vaccination) and Day 61 (post-vaccination)
Population: Analysis was performed on PPASC. Here, 'number analyzed'=participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration)
Number analyzed (Participants) | 149 | 147
titers
  Anti-Polio type 1: Day 31: number analyzed (Participants) | 147 | 146
  Anti-Polio type 1: Day 31 | 94.7 [75.5 to 119] | 109 [86.0 to 138]
  Anti-Polio type 1: Day 61 | 3135 [2692 to 3650] | 3266 [2778 to 3840]
  Anti-Polio type 2: Day 31: number analyzed (Participants) | 147 | 147
  Anti-Polio type 2: Day 31 | 227 [184 to 281] | 234 [188 to 292]
  Anti-Polio type 2: Day 61: number analyzed (Participants) | 147 | 147
  Anti-Polio type 2: Day 61 | 3344 [2635 to 4245] | 2648 [2074 to 3381]
  Anti-Polio type 3: Day 31: number analyzed (Participants) | 147 | 147
  Anti-Polio type 3: Day 31 | 135 [105 to 174] | 155 [120 to 200]
  Anti-Polio type 3: Day 61 | 7059 [5861 to 8502] | 5591 [4647 to 6728]

10. Secondary Outcome: Geometric Mean Concentrations (GMCs) of Anti-Pertussis Antibodies Contained in Tetanus, Diphtheria, and Acellular Pertussis - Inactivated Polio Vaccine (Tdap-IPV) Vaccine in Groups 1 and 2
Description: GMCs of anti-pertussis antibodies (pertussis toxoid [PT], filamentous hemagglutinin [FHA], pertactin [PRN]) and fimbriae types 2 and 3 [FIM], were measured by electro chemiluminescent method. Blood samples were assessed for participants at Day 31 and at Day 61, respectively.
Time Frame: Day 31 (post-vaccination) and Day 61 (post-vaccination)
Population: Analysis was performed on PPASC. Here, 'number analyzed'=participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: Endotoxin units per milliliter (EU/mL)
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration)
Number analyzed (Participants) | 149 | 147
Endotoxin units per milliliter (EU/mL)
  Anti-PT: Day 31: number analyzed (Participants) | 145 | 147
  Anti-PT: Day 31 | 11.9 [10.2 to 13.8] | 12.3 [10.5 to 14.4]
  Anti-PT: Day 61 | 58.4 [50.6 to 67.4] | 59.3 [51.1 to 68.8]
  Anti-FHA: Day 31: number analyzed (Participants) | 147 | 147
  Anti-FHA: Day 31 | 47.3 [40.9 to 54.7] | 58.3 [51.4 to 66.1]
  Anti-FHA: Day 61 | 177 [156 to 200] | 210 [187 to 236]
  Anti-PRN: Day 31: number analyzed (Participants) | 147 | 147
  Anti-PRN: Day 31 | 14.5 [11.2 to 18.8] | 18.2 [14.0 to 23.7]
  Anti-PRN: Day 61 | 331 [265 to 414] | 394 [316 to 491]
  Anti-FIM: Day 31: number analyzed (Participants) | 147 | 147
  Anti-FIM: Day 31 | 2.74 [2.23 to 3.37] | 3.18 [2.56 to 3.95]
  Anti-FIM: Day 61 | 152 [112 to 207] | 194 [140 to 271]

11. Secondary Outcome: Geometric Mean Concentrations (GMCs) of Anti-Diphtheria, Tetanus Antibodies Contained in Tetanus, Diphtheria, and Acellular Pertussis - Inactivated Polio Vaccine (Tdap-IPV) Vaccine: Group 3
Description: GMCs of anti-diphtheria, and tetanus antibodies were measured by electro chemiluminescent method. Blood samples were assessed for participants at Day 01 and at Day 31, respectively.
Time Frame: Day 01 (pre-vaccination) and Day 31 (post-vaccination)
Population: Analysis was performed on PPASC.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration)
Number analyzed (Participants) | 113
IU/mL
  Anti-Tetanus: Day 01 | 0.708 [0.574 to 0.874]
  Anti-Tetanus: Day 31 | 34.5 [30.1 to 39.6]
  Anti-Diphtheria: Day 01 | 0.256 [0.208 to 0.316]
  Anti-Diphtheria: Day 31 | 2.91 [2.46 to 3.44]

12. Secondary Outcome: Geometric Mean Concentrations (GMCs) of Anti-Polio Antibodies Contained in Tetanus, Diphtheria, and Acellular Pertussis - Inactivated Polio Vaccine (Tdap-IPV) Vaccine: Group 3
Description: GMCs of anti-poliovirus types 1, 2, and 3 were measured by neutralization assay. Concentrations were expressed in terms of titers (1/dilution). Blood samples were assessed for participants at Day 01 and at Day 31, respectively.
Time Frame: Day 01 (pre-vaccination) and Day 31 (post-vaccination)
Population: Analysis was performed on PPASC.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration)
Number analyzed (Participants) | 113
titers
  Anti-Polio type 1: Day 01 | 146 [112 to 190]
  Anti-Polio type 1: Day 31 | 1593 [1306 to 1943]
  Anti-Polio type 2: Day 01 | 225 [178 to 285]
  Anti-Polio type 2: Day 31 | 2950 [2409 to 3613]
  Anti-Polio type 3: Day 01 | 221 [162 to 302]
  Anti-Polio type 3: Day 31 | 3166 [2553 to 3926]

13. Secondary Outcome: Geometric Mean Concentrations (GMCs) of Anti-Pertussis Antibodies Contained in Tetanus, Diphtheria, and Acellular Pertussis - Inactivated Polio Vaccine (Tdap-IPV) Vaccine: Group 3
Description: GMCs of anti-pertussis antibodies (PT, FHA, FIM, and PRN) antibodies were measured by electro chemiluminescent method. Blood samples were assessed for participants at Day 01 and at Day 31, respectively.
Time Frame: Day 01 (pre-vaccination) and Day 31 (post-vaccination)
Population: Analysis was performed on PPASC.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration)
Number analyzed (Participants) | 113
EU/mL
  Anti-PT: Day 01 | 8.77 [7.07 to 10.9]
  Anti-PT: Day 31 | 41.4 [36.1 to 47.4]
  Anti-FHA: Day 01 | 44.5 [37.5 to 52.9]
  Anti-FHA: Day 31 | 146 [128 to 166]
  Anti-PRN: Day 01 | 11.4 [8.40 to 15.6]
  Anti-PRN: Day 31 | 236 [184 to 303]
  Anti-FIM: Day 01 | 2.32 [1.84 to 2.94]
  Anti-FIM: Day 31 | 106 [75.3 to 149]

14. Secondary Outcome: Geometric Mean Concentrations Ratios (GMCRs) of Antibodies Against Antigens Contained in Tetanus, Diphtheria, and Acellular Pertussis - Inactivated Polio Vaccine (Tdap-IPV) Vaccine in Groups 1 and 2
Description: Anti-Diphtheria, Tetanus, and Pertussis (PT, FHA, FIM, and PRN) antibodies were measured by electro chemiluminescent method. Anti-poliovirus types 1, 2, and 3 were measured by neutralization assay. GMCRs were calculated as the ratio of GMCs at Day 61 and Day 31. Blood samples were assessed for participants at Day 31 and at Day 61, respectively.
Time Frame: Day 31 (post-vaccination) and Day 61 (post-vaccination)
Population: Analysis was performed on PPASC. Here, 'number analyzed' = participants with available data for specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration)
Number analyzed (Participants) | 149 | 147
ratio
  Anti-Tetanus: number analyzed (Participants) | 147 | 147
  Anti-Tetanus | 0.677 [0.646 to 0.710] | 0.876 [0.824 to 0.931]
  Anti-Diphtheria: number analyzed (Participants) | 147 | 147
  Anti-Diphtheria | 18.5 [15.3 to 22.5] | 18.1 [15.1 to 21.7]
  Anti-Polio type 1: number analyzed (Participants) | 147 | 146
  Anti-Polio type 1 | 32.9 [24.5 to 44.2] | 29.5 [22.1 to 39.4]
  Anti-Polio type 2: number analyzed (Participants) | 145 | 147
  Anti-Polio type 2 | 14.9 [10.8 to 20.5] | 11.3 [8.09 to 15.8]
  Anti-Polio type 3: number analyzed (Participants) | 147 | 147
  Anti-Polio type 3 | 51.8 [38.0 to 70.5] | 36.1 [26.7 to 48.8]
  Anti-PT: number analyzed (Participants) | 145 | 147
  Anti-PT | 4.90 [4.36 to 5.51] | 4.83 [4.33 to 5.38]
  Anti-FHA: number analyzed (Participants) | 147 | 147
  Anti-FHA | 3.76 [3.24 to 4.35] | 3.61 [3.18 to 4.09]
  Anti-PRN: number analyzed (Participants) | 147 | 147
  Anti-PRN | 22.4 [17.9 to 27.9] | 21.6 [16.9 to 27.7]
  Anti-FIM: number analyzed (Participants) | 147 | 147
  Anti-FIM | 55.3 [44.4 to 68.9] | 61.2 [49.4 to 75.8]

15. Secondary Outcome: Geometric Mean Concentrations Ratios (GMCRs) of Antibodies Against Antigens Contained in Tetanus, Diphtheria, and Acellular Pertussis - Inactivated Polio Vaccine (Tdap-IPV) Vaccine: Group 3
Description: Anti-Diphtheria, Tetanus, and Pertussis (PT, FHA, FIM, and PRN) antibodies were measured by electro chemiluminescent method. Anti-poliovirus types 1, 2, and 3 were measured by neutralization assay. GMCRs were calculated as the ratio of GMCs at Day 31/Day 01. Blood samples were assessed for participants at Day 01 and at Day 31, respectively.
Time Frame: Day 01 (pre-vaccination) and Day 31 (post-vaccination)
Population: Analysis was performed on PPASC.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration)
Number analyzed (Participants) | 113
ratio
  Anti-Tetanus | 48.7 [40.1 to 59.3]
  Anti-Diphtheria | 11.4 [9.17 to 14.1]
  Anti-Polio type 1 | 10.9 [7.77 to 15.4]
  Anti-Polio type 2 | 13.1 [9.66 to 17.8]
  Anti-Polio type 3 | 14.3 [10.1 to 20.3]
  Anti-PT | 4.72 [4.05 to 5.49]
  Anti-FHA | 3.27 [2.82 to 3.80]
  Anti-PRN | 20.6 [15.7 to 27.1]
  Anti-FIM | 45.7 [35.7 to 58.5]

16. Secondary Outcome: Percentage of Participants With Antibody Titers Above Predefined Thresholds Against Antigens Contained in Tetanus, Diphtheria, and Acellular Pertussis - Inactivated Polio Vaccine (Tdap-IPV) Vaccine in Groups 1 and 2
Description: Antibody titers above predefined thresholds against Tdap-IPV vaccine antigens were defined as: Anti-D Ab titers and Anti-T Ab titers >= 0.1 IU/mL, and >= 1.0 IU/mL; Anti-Polio 1, 2, and 3 Ab titers >= 8 (1/dilution). Blood samples were assessed for participants at Day 31 and at Day 61, respectively.
Time Frame: Day 31 (post-vaccination) and Day 61 (post-vaccination)
Population: Analysis was performed on PPASC. Here, 'number analyzed' = participants with available data for specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration)
Number analyzed (Participants) | 149 | 147
percentage of participants
  Anti-T: Day 31: >=0.1: number analyzed (Participants) | 147 | 147
  Anti-T: Day 31: >=0.1 | 100 [97.5 to 100] | 100 [97.5 to 100]
  Anti-T: Day 31: >=1.0: number analyzed (Participants) | 147 | 147
  Anti-T: Day 31: >=1.0 | 100 [97.5 to 100] | 98.0 [94.2 to 99.6]
  Anti-T: Day 61: >=0.1 | 100 [97.6 to 100] | 100 [97.5 to 100]
  Anti-T: Day 61: >=1.0 | 99.3 [96.3 to 100] | 100 [97.5 to 100]
  Anti-D: Day 31: >=0.1: number analyzed (Participants) | 147 | 147
  Anti-D: Day 31: >=0.1 | 76.9 [69.2 to 83.4] | 79.6 [72.2 to 85.8]
  Anti-D: Day 31: >=1.0: number analyzed (Participants) | 147 | 147
  Anti-D: Day 31: >=1.0 | 4.8 [1.9 to 9.6] | 4.8 [1.9 to 9.6]
  Anti-D: Day 61: >=0.1 | 100 [97.6 to 100] | 100 [97.5 to 100]
  Anti-D: Day 61: >=1.0 | 93.3 [88.0 to 96.7] | 92.5 [87.0 to 96.2]
  Anti-Polio 1: Day 31: >=8: number analyzed (Participants) | 147 | 146
  Anti-Polio 1: Day 31: >=8 | 95.2 [90.4 to 98.1] | 95.2 [90.4 to 98.1]
  Anti-Polio 1: Day 61: >=8 | 100 [97.6 to 100] | 100 [97.5 to 100]
  Anti-Polio 2: Day 31: >=8: number analyzed (Participants) | 147 | 147
  Anti-Polio 2: Day 31: >=8 | 99.3 [96.3 to 100] | 100 [97.5 to 100]
  Anti-Polio 2: Day 61: >=8: number analyzed (Participants) | 147 | 147
  Anti-Polio 2: Day 61: >=8 | 100 [97.5 to 100] | 100 [97.5 to 100]
  Anti-Polio 3: Day 31: >=8: number analyzed (Participants) | 147 | 147
  Anti-Polio 3: Day 31: >=8 | 95.9 [91.3 to 98.5] | 96.6 [92.2 to 98.9]
  Anti-Polio 3: Day 61: >=8 | 100 [97.6 to 100] | 100 [97.5 to 100]

17. Secondary Outcome: Percentage of Participants With Antibody Titers Above Predefined Thresholds Against Antigens Contained in Tetanus, Diphtheria, and Acellular Pertussis - Inactivated Polio Vaccine (Tdap-IPV) Vaccine: Group 3
Description: Antibody titers above predefined thresholds against Tdap-IPV vaccine antigens were defined as: Anti-D Ab titers and Anti-T Ab titers >= 0.1 IU/mL, and >= 1.0 IU/mL; Anti-Polio 1, 2, and 3 Ab titers >= 8 (1/dilution). Blood samples were assessed for participants at Day 01 and at Day 31, respectively.
Time Frame: Day 01 (pre-vaccination) and Day 31 (post-vaccination)
Population: Analysis was performed on PPASC.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration)
Number analyzed (Participants) | 113
percentage of participants
  Anti-T: Day 01: >=0.1 | 96.5 [91.2 to 99.0]
  Anti-T: Day 01: >=1.0 | 38.9 [29.9 to 48.6]
  Anti-T: Day 31: >=0.1 | 100 [96.8 to 100]
  Anti-T: Day 31: >=1.0 | 100 [96.8 to 100]
  Anti-D: Day 01: >=0.1 | 85.0 [77.0 to 91.0]
  Anti-D: Day 01: >=1.0 | 9.7 [5.0 to 16.8]
  Anti-D: Day 31: >=0.1 | 99.1 [95.2 to 100]
  Anti-D: Day 31: >=1.0 | 90.3 [83.2 to 95.0]
  Anti-Polio 1: Day 01: >=8 | 99.1 [95.2 to 100]
  Anti-Polio 1: Day 31: >=8 | 100 [96.8 to 100]
  Anti-Polio 2: Day 01: >=8 | 100 [96.8 to 100]
  Anti-Polio 2: Day 31: >=8 | 100 [96.8 to 100]
  Anti-Polio 3: Day 01: >=8 | 96.5 [91.2 to 99.0]
  Anti-Polio 3: Day 31: >=8 | 100 [96.8 to 100]

18. Secondary Outcome: Percentage of Participants With Vaccine Seroresponse Against Pertussis Antigens
Description: Vaccine seroresponse was defined as post-vaccination concentration >= 4 * Baseline concentration, if the anti-pertussis antibody concentration at Baseline was < 4*lower limit of quantification (LLOQ), or >= 2*Baseline concentration, if the anti-pertussis antibody concentration at Baseline was >= 4*LLOQ. Post vaccine seroresponse for anti-pertussis antigens was Day 31 for Group 3 and Day 61 for Groups 1 and 2.
Time Frame: Day 61 (post-vaccination for Groups 1 and 2) and Day 31 (post-vaccination for Group 3)
Population: Analysis was performed on PPASC. Here, 'number analyzed'=participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration)
Number analyzed (Participants) | 149 | 147 | 113
percentage of participants
  Anti-PT: number analyzed (Participants) | 145 | 147 | 113
  Anti-PT | 81.4 [74.1 to 87.4] | 83.0 [75.9 to 88.7] | 76.1 [67.2 to 83.6]
  Anti-FHA: number analyzed (Participants) | 147 | 147 | 113
  Anti-FHA | 74.8 [67.0 to 81.6] | 76.2 [68.5 to 82.8] | 70.8 [61.5 to 79.0]
  Anti-PRN: number analyzed (Participants) | 147 | 147 | 113
  Anti-PRN | 98.0 [94.2 to 99.6] | 94.6 [89.6 to 97.6] | 91.2 [84.3 to 95.7]
  Anti-FIM: number analyzed (Participants) | 147 | 147 | 113
  Anti-FIM | 93.9 [88.7 to 97.2] | 97.3 [93.2 to 99.3] | 95.6 [90.0 to 98.5]

19. Secondary Outcome: Geometric Mean Titers (GMTs) of Antibodies Against Antigens Contained in Human Papillomavirus (HPV) Vaccine in Groups 1 and 2
Description: Anti-HPV antibodies were measured by the direct virus-like particle (VLP) electrochemiluminescence multi-plex immunoassay for detection of antibodies towards HPV types 6, 11, 16, 18, 31, 33, 45, 52, and 58. Titers were expressed in terms of 1/dilution. Blood samples were assessed for participants at Day 31 and at Day 61, respectively.
Time Frame: Day 31 (post-vaccination) and Day 61 (post-vaccination)
Population: Analysis was performed on PPASC. Here, 'number analyzed'=participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration)
Number analyzed (Participants) | 149 | 147
titers
  Anti-HPV type-6: Day 31: number analyzed (Participants) | 147 | 147
  Anti-HPV type-6: Day 31 | 2.30 [1.94 to 2.73] | 2.03 [1.74 to 2.37]
  Anti-HPV type-6: Day 61 | 73.9 [64.3 to 85.0] | 64.8 [55.8 to 75.4]
  Anti-HPV type-11: Day 31: number analyzed (Participants) | 147 | 147
  Anti-HPV type-11: Day 31 | 1.11 [1.05 to 1.18] | 1.08 [1.03 to 1.13]
  Anti-HPV type-11: Day 61 | 43.9 [38.9 to 49.5] | 39.3 [33.9 to 45.5]
  Anti-HPV type-16: Day 31: number analyzed (Participants) | 147 | 147
  Anti-HPV type-16: Day 31 | 2.06 [1.95 to 2.17] | 2.08 [1.97 to 2.19]
  Anti-HPV type-16: Day 61 | 199 [171 to 231] | 168 [142 to 199]
  Anti-HPV type-18: Day 31: number analyzed (Participants) | 147 | 147
  Anti-HPV type-18: Day 31 | 1.59 [1.50 to 1.70] | 1.52 [1.49 to 1.54]
  Anti-HPV type-18: Day 61 | 46.5 [38.4 to 56.4] | 38.5 [31.3 to 47.4]
  Anti-HPV type-31: Day 31: number analyzed (Participants) | 147 | 147
  Anti-HPV type-31: Day 31 | 1.08 [0.995 to 1.18] | 1.05 [1.01 to 1.10]
  Anti-HPV type-31: Day 61 | 31.7 [26.5 to 38.1] | 28.9 [24.0 to 34.9]
  Anti-HPV type-33: Day 31: number analyzed (Participants) | 147 | 147
  Anti-HPV type-33: Day 31 | 1.01 [0.987 to 1.04] | 1.02 [0.997 to 1.04]
  Anti-HPV type-33: Day 61 | 21.1 [17.8 to 24.9] | 19.1 [16.1 to 22.7]
  Anti-HPV type-45: Day 31: number analyzed (Participants) | 147 | 147
  Anti-HPV type-45: Day 31 | 0.520 [0.499 to 0.543] | 0.509 [0.492 to 0.527]
  Anti-HPV type-45: Day 61 | 11.5 [9.35 to 14.1] | 9.54 [7.68 to 11.9]
  Anti-HPV type-52: Day 31: number analyzed (Participants) | 147 | 147
  Anti-HPV type-52: Day 31 | 0.535 [0.503 to 0.569] | 0.514 [0.498 to 0.530]
  Anti-HPV type-52: Day 61 | 47.4 [41.1 to 54.7] | 39.3 [33.5 to 46.1]
  Anti-HPV type-58: Day 31: number analyzed (Participants) | 147 | 147
  Anti-HPV type-58: Day 31 | 1.09 [1.02 to 1.16] | 1.05 [1.00 to 1.10]
  Anti-HPV type-58: Day 61 | 29.6 [25.5 to 34.3] | 26.0 [22.2 to 30.4]

20. Secondary Outcome: Geometric Mean Titers (GMTs) of Antibodies Against Antigens Contained in Human Papillomavirus (HPV) Vaccine: Group 3
Description: Anti-HPV antibodies were measured by the direct VLP electrochemiluminescence multi-plex immunoassay for detection of antibodies towards HPV types 6, 11, 16, 18, 31, 33, 45, 52, and 58. Titers were expressed in terms of 1/dilution. Blood samples were assessed for participants at Day 01 and at Day 31, respectively.
Time Frame: Day 01 (pre-vaccination) and Day 31 (post-vaccination)
Population: Analysis was performed on PPASC.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration)
Number analyzed (Participants) | 113
titers
  Anti-HPV type-6: Day 01 | 2.12 [1.76 to 2.55]
  Anti-HPV type-6: Day 31 | 50.6 [42.0 to 60.9]
  Anti-HPV type-11: Day 01 | 1.07 [1.02 to 1.13]
  Anti-HPV type-11: Day 31 | 36.3 [30.8 to 42.8]
  Anti-HPV type-16: Day 01 | 2.02 [1.98 to 2.07]
  Anti-HPV type-16: Day 31 | 146 [118 to 179]
  Anti-HPV type-18: Day 01 | 1.50 [NA to NA] — The 95% CI was not computable as the standard deviation of the sample was 0, since all participants had the same value.
  Anti-HPV type-18: Day 31 | 31.2 [24.0 to 40.6]
  Anti-HPV type-31: Day 01 | 1.07 [1.02 to 1.13]
  Anti-HPV type-31: Day 31 | 24.7 [19.2 to 31.8]
  Anti-HPV type-33: Day 01 | 1.01 [0.989 to 1.03]
  Anti-HPV type-33: Day 31 | 15.0 [12.2 to 18.6]
  Anti-HPV type-45: Day 01 | 0.524 [0.493 to 0.556]
  Anti-HPV type-45: Day 31 | 8.24 [6.30 to 10.8]
  Anti-HPV type-52: Day 01 | 0.521 [0.500 to 0.544]
  Anti-HPV type-52: Day 31 | 40.9 [33.5 to 49.8]
  Anti-HPV type-58: Day 01 | 1.08 [1.02 to 1.14]
  Anti-HPV type-58: Day 31 | 20.6 [16.9 to 25.1]

21. Secondary Outcome: Geometric Mean Titers Ratios (GMTRs) of Antibodies Against Antigens Contained in Human Papillomavirus (HPV) Vaccine in Groups 1 and 2
Description: Anti-HPV antibodies were measured by the direct virus-like particle (VLP) electrochemiluminescence multi-plex immunoassay for detection of antibodies towards HPV types 6, 11, 16, 18, 31, 33, 45, 52, and 58. GMTRs were calculated as the ratio of GMTs at Day 61/Day 31. Blood samples were assessed for participants at Day 31 and at Day 61, respectively.
Time Frame: Day 31 (post-vaccination) and Day 61 (post-vaccination)
Population: Analysis was performed on PPASC. Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration)
Number analyzed (Participants) | 147 | 147
ratio
  Anti-HPV type-6 | 32.0 [26.5 to 38.6] | 31.9 [26.5 to 38.5]
  Anti-HPV type-11 | 39.0 [34.2 to 44.5] | 36.5 [31.3 to 42.7]
  Anti-HPV type-16 | 96.6 [83.4 to 112] | 80.8 [68.1 to 95.8]
  Anti-HPV type-18 | 29.7 [24.4 to 36.2] | 25.4 [20.6 to 31.2]
  Anti-HPV type-31 | 29.8 [25.1 to 35.4] | 27.5 [22.8 to 33.2]
  Anti-HPV type-33 | 20.8 [17.7 to 24.4] | 18.7 [15.8 to 22.2]
  Anti-HPV type-45 | 21.9 [17.9 to 26.9] | 18.8 [15.1 to 23.3]
  Anti-HPV type-52 | 88.0 [77.1 to 100] | 76.5 [65.0 to 90.1]
  Anti-HPV type-58 | 27.1 [23.3 to 31.4] | 24.8 [21.2 to 29.0]

22. Secondary Outcome: Geometric Mean Titers Ratios (GMTRs) of Antibodies Against Antigens Contained in Human Papillomavirus (HPV) Vaccine: Group 3
Description: Anti-HPV antibodies were measured by the direct VLP electrochemiluminescence multi-plex immunoassay for detection of antibodies towards HPV types 6, 11, 16, 18, 31, 33, 45, 52, and 58. GMTRs were calculated as the ratio of GMTs at Day 31/Day 01. Blood samples were assessed for participants at Day 01 and at Day 31, respectively.
Time Frame: Day 01 (pre-vaccination) and Day 31 (post-vaccination)
Population: Analysis was performed on PPASC.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration)
Number analyzed (Participants) | 113
ratio
  Anti-HPV type-6 | 23.9 [19.4 to 29.3]
  Anti-HPV type-11 | 33.9 [28.6 to 40.1]
  Anti-HPV type-16 | 71.9 [58.6 to 88.2]
  Anti-HPV type-18 | 20.8 [16.0 to 27.1]
  Anti-HPV type-31 | 23.1 [17.9 to 29.6]
  Anti-HPV type-33 | 14.9 [12.0 to 18.4]
  Anti-HPV type-45 | 15.7 [12.0 to 20.7]
  Anti-HPV type-52 | 78.4 [64.3 to 95.5]
  Anti-HPV type-58 | 19.1 [15.8 to 23.2]

23. Secondary Outcome: Percentage of Participants With Vaccine Seroconversion Against Antigens Contained in Human Papillomavirus (HPV) Vaccine
Description: Vaccine Seroconversion was defined as changing serostatus from seronegative (participants with a titer inferior to the serostatus cut-off value) at Baseline to seropositive after vaccination. A participant with a titer at or above the serostatus cut-off for a given HPV type was considered seropositive for that type. The serostatus cut-offs for HPV types 6, 11, 16, 18, 31, 33, 45, 52, and 58 were 9, 6, 5, 5, 3, 4, 3, 5 and 5 milli-Merck units (mMU)/mL, respectively. Post vaccine seroconversion for antigens contained in HPV vaccine was Day 31 for Group 3 and Day 61 for Groups 1 and 2.
Time Frame: Day 61 (post-vaccination for Groups 1 and 2) and Day 31 (post-vaccination for Group 3)
Population: Analysis was performed on PPASC. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration)
Number analyzed (Participants) | 147 | 147 | 113
percentage of participants
  Anti-HPV type-6 | 87.8 [81.3 to 92.6] | 88.4 [82.1 to 93.1] | 85.0 [77.0 to 91.0]
  Anti-HPV type-11 | 99.3 [96.3 to 100] | 97.3 [93.2 to 99.3] | 97.3 [92.4 to 99.4]
  Anti-HPV type-16 | 99.3 [96.3 to 100] | 96.6 [92.2 to 98.9] | 98.2 [93.8 to 99.8]
  Anti-HPV type-18 | 94.6 [89.6 to 97.6] | 92.5 [87.0 to 96.2] | 88.5 [81.1 to 93.7]
  Anti-HPV type-31 | 96.6 [92.2 to 98.9] | 93.2 [87.8 to 96.7] | 88.5 [81.1 to 93.7]
  Anti-HPV type-33 | 95.2 [90.4 to 98.1] | 91.8 [86.2 to 95.7] | 87.6 [80.1 to 93.1]
  Anti-HPV type-45 | 81.6 [74.4 to 87.5] | 83.0 [75.9 to 88.7] | 75.2 [66.2 to 82.9]
  Anti-HPV type-52 | 99.3 [96.3 to 100] | 98.0 [94.2 to 99.6] | 96.5 [91.2 to 99.0]
  Anti-HPV type-58 | 95.2 [90.4 to 98.1] | 92.5 [87.0 to 96.2] | 92.0 [85.4 to 96.3]

24. Secondary Outcome: Number of Participants Reporting Immediate Unsolicited Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a patient or in a clinical investigation participant administered a medicinal product and which did not had any casual relationship with the treatment. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the case report form (CRF) in terms of diagnosis and/or onset window post-vaccination. All participants were observed for 30 minutes after vaccination, and any unsolicited AEs occurred during that time were recorded as immediate unsolicited AEs in the CRB. Reported AEs for each arm were presented as pre-specified in the study protocol.
Time Frame: Within 30 minutes post-any and each vaccination (Vaccination 1 [i.e., at Day 1] and 2 [i.e., at Day 31])
Population: Analysis was performed on safety analysis set that included all participants who had received at least one dose of the study vaccines and had any safety data available. Here, 'number analyzed' = participants with available data for each specified category and "0" in the number analyzed field signifies that at Day 31, participants of Group 3 received no vaccination and thus data were not collected and analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration)
Number analyzed (Participants) | 171 | 171 | 116
Participants
  Post-any vaccination | 0 | 0 | 0
  Post-vaccination 1 | 0 | 0 | 0
  Post-vaccination 2: number analyzed (Participants) | 169 | 168 | 0
  Post-vaccination 2 | 0 | 0 |

25. Secondary Outcome: Number of Participants Reporting Solicited Injection Site Reactions
Description: SR: expected AR (sign or symptom) observed & reported under conditions (nature & onset) prelisted (i.e., solicited) in CRF & considered as related to product. Injection site reactions: pain, erythema, & swelling. Here, "0" in number analyzed for MenACYW categories signifies no participant were evaluable as in Group (Gps.) 2 MenACYW vaccine was not administered; for Gps.1& 3: "0" in number analyzed for Nimenrix signifies no participant were evaluable as in Gps. 1 & 3 Nimenrix was not administered. At Vaccination (vacc.)1 (Gps.1 & 2): "0" in number analyzed for 9vHPV & Tadp-IPV signifies no participant were evaluable as these vaccines were not administered at vacc.1 (Day01). At Vacc. 2 (Gps.1, 2 & 3): "0" in number analyzed for MenACYW and Nimenrix signifies no participant were evaluable as these vaccines were not administered at vacc. 2 (Day 31); & for Gps. 3 "0" in number analyzed for 9vHPV and Tadp-IPV signifies no participant were evaluable as these vaccines were not administered.
Time Frame: Within 7 days post-any and each vaccination (Vaccination 1 [i.e., at Day 1] and 2 [i.e., at Day 31])
Population: Analysis was performed on safety analysis set. Here, 'Number analyzed'=participants with available data for specified category. The assessment of injection site reactions (pain, swelling and erythema) after the MenACYW Conjugate vaccines (MenQuadfi and Nimenrix) and 2 other adolescent vaccines allowed in the assessment of local reactogenicity and helped in identifying injection site reaction per vaccine received. Reported AEs for each arm were presented as pre-specified in the study protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccine (Sequential Administration): Participants received 0.5 mL intramuscular injection of Nimenrix® vaccine on Day 01 and 0.5-mL intramuscular injection of 9vHPV + Tdap-IPV vaccines (sequentially after Nimenrix® vaccine) at Day 31.
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccine (Sequential Administration) | Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration)
Number analyzed (Participants) | 171 | 171 | 116
Participants
  MenACYW Conjugate vaccine: Pain: Post-any vaccination: number analyzed (Participants) | 169 | 0 | 116
  MenACYW Conjugate vaccine: Pain: Post-any vaccination | 91 |  | 69
  MenACYW Conjugate vaccine: Erythema: Post-any vaccination: number analyzed (Participants) | 169 | 0 | 116
  MenACYW Conjugate vaccine: Erythema: Post-any vaccination | 19 |  | 11
  MenACYW Conjugate vaccine: Swelling: Post-any vaccination: number analyzed (Participants) | 169 | 0 | 116
  MenACYW Conjugate vaccine: Swelling: Post-any vaccination | 17 |  | 12
  Nimenrix vaccine: Pain: Post-any vaccination: number analyzed (Participants) | 0 | 170 | 0
  Nimenrix vaccine: Pain: Post-any vaccination |  | 87 |
  Nimenrix vaccine: Erythema: Post-any vaccination: number analyzed (Participants) | 0 | 170 | 0
  Nimenrix vaccine: Erythema: Post-any vaccination |  | 3 |
  Nimenrix vaccine: Swelling: Post-any vaccination: number analyzed (Participants) | 0 | 170 | 0
  Nimenrix vaccine: Swelling: Post-any vaccination |  | 7 |
  9vHPV: Pain: Post-any vaccination: number analyzed (Participants) | 168 | 165 | 116
  9vHPV: Pain: Post-any vaccination | 113 | 125 | 97
  9vHPV: Erythema: Post-any vaccination: number analyzed (Participants) | 168 | 165 | 116
  9vHPV: Erythema: Post-any vaccination | 7 | 3 | 6
  9vHPV: Swelling: Post-any vaccination: number analyzed (Participants) | 168 | 165 | 116
  9vHPV: Swelling: Post-any vaccination | 4 | 3 | 7
  Tdap-IPV: Pain: Post-any vaccination: number analyzed (Participants) | 168 | 164 | 116
  Tdap-IPV: Pain: Post-any vaccination | 116 | 117 | 95
  Tdap-IPV: Erythema: Post-any vaccination: number analyzed (Participants) | 168 | 164 | 116
  Tdap-IPV: Erythema: Post-any vaccination | 9 | 5 | 13
  Tdap-IPV: Swelling: Post-any vaccination: number analyzed (Participants) | 168 | 164 | 116
  Tdap-IPV: Swelling: Post-any vaccination | 9 | 3 | 10
  MenACYW Conjugate vaccine: Pain: Post-vaccination 1: number analyzed (Participants) | 169 | 0 | 116
  MenACYW Conjugate vaccine: Pain: Post-vaccination 1 | 91 |  | 69
  MenACYW Conjugate vaccine: Erythema: Post-vaccination 1: number analyzed (Participants) | 169 | 0 | 116
  MenACYW Conjugate vaccine: Erythema: Post-vaccination 1 | 19 |  | 11
  MenACYW Conjugate vaccine: Swelling: Post-vaccination 1: number analyzed (Participants) | 169 | 0 | 116
  MenACYW Conjugate vaccine: Swelling: Post-vaccination 1 | 17 |  | 12
  Nimenrix vaccine: Pain: Post-vaccination 1: number analyzed (Participants) | 0 | 170 | 0
  Nimenrix vaccine: Pain: Post-vaccination 1 |  | 87 |
  Nimenrix vaccine: Erythema: Post-vaccination 1: number analyzed (Participants) | 0 | 170 | 0
  Nimenrix vaccine: Erythema: Post-vaccination 1 |  | 3 |
  Nimenrix vaccine: Swelling: Post-vaccination 1: number analyzed (Participants) | 0 | 170 | 0
  Nimenrix vaccine: Swelling: Post-vaccination 1 |  | 7 |
  9vHPV: Pain: Post-vaccination 1: number analyzed (Participants) | 0 | 0 | 116
  9vHPV: Pain: Post-vaccination 1 |  |  | 97
  9vHPV: Erythema: Post-vaccination 1: number analyzed (Participants) | 0 | 0 | 116
  9vHPV: Erythema: Post-vaccination 1 |  |  | 6
  9vHPV: Swelling: Post-vaccination 1: number analyzed (Participants) | 0 | 0 | 116
  9vHPV: Swelling: Post-vaccination 1 |  |  | 7
  Tdap-IPV: Pain: Post-vaccination 1: number analyzed (Participants) | 0 | 0 | 116
  Tdap-IPV: Pain: Post-vaccination 1 |  |  | 95
  Tdap-IPV: Erythema: Post-vaccination 1: number analyzed (Participants) | 0 | 0 | 116
  Tdap-IPV: Erythema: Post-vaccination 1 |  |  | 13
  Tdap-IPV: Swelling: Post-vaccination 1: number analyzed (Participants) | 0 | 0 | 116
  Tdap-IPV: Swelling: Post-vaccination 1 |  |  | 10
  MenACYW Conjugate vaccine: Pain: Post-vaccination 2: number analyzed (Participants) | 0 | 0 | 0
  MenACYW Conjugate vaccine: Erythema: Post-vaccination 2: number analyzed (Participants) | 0 | 0 | 0
  MenACYW Conjugate vaccine: Swelling: Post-vaccination 2: number analyzed (Participants) | 0 | 0 | 0
  Nimenrix vaccine: Pain: Post-vaccination 2: number analyzed (Participants) | 0 | 0 | 0
  Nimenrix vaccine: Erythema: Post-vaccination 2: number analyzed (Participants) | 0 | 0 | 0
  Nimenrix vaccine: Swelling: Post-vaccination 2: number analyzed (Participants) | 0 | 0 | 0
  9vHPV: Pain: Post-vaccination 2: number analyzed (Participants) | 168 | 165 | 0
  9vHPV: Pain: Post-vaccination 2 | 113 | 125 |
  9vHPV: Erythema: Post-vaccination 2: number analyzed (Participants) | 168 | 165 | 0
  9vHPV: Erythema: Post-vaccination 2 | 7 | 3 |
  9vHPV: Swelling: Post-vaccination 2: number analyzed (Participants) | 168 | 165 | 0
  9vHPV: Swelling: Post-vaccination 2 | 4 | 3 |
  Tdap-IPV: Pain: Post-vaccination 2: number analyzed (Participants) | 168 | 164 | 0
  Tdap-IPV: Pain: Post-vaccination 2 | 116 | 117 |
  Tdap-IPV: Erythema: Post-vaccination 2: number analyzed (Participants) | 168 | 164 | 0
  Tdap-IPV: Erythema: Post-vaccination 2 | 9 | 5 |
  Tdap-IPV: Swelling: Post-vaccination 2: number analyzed (Participants) | 168 | 164 | 0
  Tdap-IPV: Swelling: Post-vaccination 2 | 9 | 3 |

26. Secondary Outcome: Number of Participants Reporting Solicited Systemic Reactions
Description: A solicited reaction (SR) was an expected adverse reaction (AR) (sign or symptom) observed and reported under the conditions (nature and onset) prelisted (i.e., solicited) in the CRF and considered as related to the product administered. Solicited systemic reactions included fever, headache, malaise, and myalgia. Reported AEs for each arm were presented as pre-specified in the study protocol.
Time Frame: Within 7 days post-any and each vaccination (Vaccination 1 [i.e., at Day 1] and 2 [i.e., at Day 31])
Population: Analysis was performed on safety analysis set. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category and "0" in the number analyzed field signifies that at Day 31, participants of Group 3 received no vaccination and thus data were not collected and analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration)
Number analyzed (Participants) | 169 | 170 | 116
Participants
  Fever: Post-any vaccination | 12 | 11 | 6
  Headache: Post-any vaccination | 75 | 64 | 52
  Malaise: Post-any vaccination | 65 | 48 | 42
  Myalgia: Post-any vaccination | 84 | 81 | 67
  Fever: Post-vaccination 1 | 7 | 4 | 6
  Headache: Post-vaccination 1: number analyzed (Participants) | 168 | 170 | 116
  Headache: Post-vaccination 1 | 59 | 44 | 52
  Malaise: Post-vaccination 1 | 46 | 32 | 42
  Myalgia: Post-vaccination 1 | 51 | 53 | 67
  Fever: Post-vaccination 2: number analyzed (Participants) | 168 | 165 | 0
  Fever: Post-vaccination 2 | 6 | 7 |
  Headache: Post-vaccination 2: number analyzed (Participants) | 168 | 165 | 0
  Headache: Post-vaccination 2 | 37 | 40 |
  Malaise: Post-vaccination 2: number analyzed (Participants) | 168 | 165 | 0
  Malaise: Post-vaccination 2 | 40 | 26 |
  Myalgia: Post-vaccination 2: number analyzed (Participants) | 168 | 165 | 0
  Myalgia: Post-vaccination 2 | 67 | 61 |

27. Secondary Outcome: Number of Participants Reporting Unsolicited Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a patient or in a clinical investigation participant administered a medicinal product and which did not had any casual relationship with the treatment. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the case report book (CRB) in terms of diagnosis and/or onset window post-vaccination. Reported AEs for each arm were presented as pre-specified in the study protocol.
Time Frame: From Day 01 up to Day 31 post-any and each vaccination (Vaccination 1 [i.e., at Day 1] and 2 [i.e., at Day 31])
Population: Analysis was performed on safety analysis set. Here, 'Number analyzed' = participants with available data for each specified category and "0" in the number analyzed field signifies that at Day 31, participants of Group 3 received no vaccination and thus data were not collected and analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration)
Number analyzed (Participants) | 171 | 171 | 116
Participants
  Post-any vaccination | 69 | 49 | 37
  Post-vaccination 1 | 49 | 31 | 37
  Post-vaccination 2: number analyzed (Participants) | 169 | 168 | 0
  Post-vaccination 2 | 34 | 27 |

28. Secondary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs) Including Adverse Events of Special Interest (AESI)
Description: A SAE was any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. A SAE which caused death of the participant was considered as fatal SAE. Adverse events of special interest (AESIs) were defined as event for which ongoing monitoring and rapid communication by the investigator to the sponsor was done. Reported AEs for each arm were presented as pre-specified in the study protocol.
Time Frame: From Day 01 up to the last study day (i.e., Day 61 for Groups 1 and 2 and Day 31 for Group 3)
Population: Analysis was performed on safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration)
Number analyzed (Participants) | 171 | 171 | 116
Participants
  SAE | 0 | 1 | 0
  AESI | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Unsolicited AE data were collected from Day 01 up to Day 31 post-any vaccination. Solicited reaction data were collected from Day 01 up to Day 7 post-any vaccination. The SAEs were collected up to the last study day i.e., Day 61 for Groups 1 and 2 and Day 31 for Group 3
Description: SR was an expected AR that was prelisted (i.e., solicited) in the CRF and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the CRF (i.e., solicited) in terms of symptom and/or onset post-vaccination. Analysis was performed on safety analysis set. In AE section, solicited reaction Fever is reported under Pyrexia. Reported AEs for each arm were presented as pre-specified in study protocol.
Arm/Group | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) | Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration)
All-Cause Mortality (participants affected / at risk) | 0/171 | 0/171 | 0/116
Serious Adverse Events (participants affected / at risk) | 0/171 | 1/171 | 0/116
Other Adverse Events (participants affected / at risk) | 153/171 | 151/171 | 112/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) (N=171) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) (N=171) | Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration) (N=116)
Type 1 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) (N=171) | Group 2: Nimenrix® + 9vHPV + Tdap-IPV Vaccines (Sequential Administration) (N=171) | Group 3: MenACYW Conjugate Vaccine + 9vHPV + Tdap-IPV Vaccines (Concomitant Administration) (N=116)
Injection Site Bruising (General disorders) | 7 (8) | 9 (10) | 3 (3)
Injection Site Erythema (General disorders) | 27 (35) | 9 (11) | 18 (30)
Injection Site Pain (General disorders) | 144 (320) | 140 (329) | 107 (261)
Injection Site Swelling (General disorders) | 25 (30) | 13 (13) | 15 (30)
Malaise (General disorders) | 65 (86) | 48 (58) | 42 (42)
Pyrexia (General disorders) | 14 (15) | 11 (11) | 6 (6) — Pyrexia/Fever events that occurred after 7 days post-vaccination were considered as unsolicited AE.
Covid-19 (Infections and infestations) | 9 (9) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 84 (118) | 81 (114) | 67 (67)
Headache (Nervous system disorders) | 76 (98) | 66 (87) | 52 (52) — Headache events that occurred after 7 days post-vaccination were considered as unsolicited AE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT04490018/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT04490018/SAP_001.pdf